CLINICAL TRIAL: NCT06731972
Title: The Impact of Using Mobile Games on Rehabilitation Outcomes in Thumb Rehabilitation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kirsehir Ahi Evran Universitesi (Other)
Responsible Party: Principal Investigator, seher karaçam, Research Assistant, MSc., Physiotherapist, Kirsehir Ahi Evran Universitesi
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 167638
Record Dates: First submitted 2024-12-02; First posted 2024-12-13 (Actual); Last update posted 2024-12-13 (Actual); Status verified 2024-12

CONDITIONS: Thumb Injury; Rehabilitation Outcome; Mobile Phone Use
Keywords: Thumb; Rehabilitation; Games; Technology
MeSH Terms: conditions — Cell Phone Use | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Routine treatment) (Active Comparator): Routine treatment (classical massage, stretching, functional exercises, electrical modalities, thermal agents, home exercises, etc.) will be applied.
  Interventions: Other: Exercises
- Group 2 (Routine treatment + mobile game) (Experimental): The routine treatment plus mobile game group will receive routine treatment along with 20-30 minutes of mobile application games (such as Temple Run, Flappy Bird, Angry Birds, etc.) daily as part of their home exercise program.
  Interventions: Other: Exercises; Device: Mobile game

INTERVENTIONS:
Other: Exercises — Classical massage, stretching, functional exercises, electrical modalities, thermal agents, home exercises, etc., plus home exercises.
Device: Mobile game — mobile application games (such as Temple Run, Flappy Bird, Angry Birds, etc., or games the patient is already playing) as part of their home exercise program.
  Arms: Group 2 (Routine treatment + mobile game)

SUMMARY:
Hand injuries and diseases are common reasons for hospital visits and lead to both functional and workforce losses, making them a persistent problem in treatment and rehabilitation approaches. Among the various functions of the hand, the thumb is of particular importance due to its large representation in the brain and its contribution to all gripping and holding functions. Loss of function in the thumb leads to a loss of at least 40% of hand skills. Therefore, restoring the thumb's original functionality is this study primary goal in rehabilitation. To achieve this goal, intensive rehabilitation is required, which cannot be fully accomplished through clinic sessions alone, as home exercises contribute significantly to this process. The low adherence of patients to home exercises has led researchers to explore various alternatives.

The aim of this study is to investigate the effect of mobile application games on rehabilitation outcomes in patients who have lost thumb function. For the pre- and post-treatment evaluations of the patients, the following assessment tools will be used: the Visual Analog Scale (VAS) for pain, the eight-shaped tape measure for edema, the Quick-DASH (Disabilities of the Arm, Shoulder, and Hand) scale for upper extremity functionality, a finger goniometer for joint range of motion, the DuruÖz Hand Index for measuring activities of daily living, and a home exercise adherence tracking form to evaluate adherence to home exercises.

As determined by this study power analysis, 38 patients with thumb injuries will be included in the study. These patients will be randomly assigned into two groups: the routine treatment group (19 patients) and the routine treatment plus mobile game group (19 patients). The routine treatment group will receive standard treatment at the Kırşehir Ahi Evran University Faculty of Physiotherapy and Rehabilitation Hand Clinic, including classical massage, stretching, functional exercises, electrical modalities, thermal agents, and home exercises. In the routine treatment plus mobile game group, in addition to the standard treatment, patients will engage in 20-30 minutes of mobile application games (e.g., Temple Run, Flappy Bird, Angry Birds) as part of their home exercise program.

Researchers hypothesize that the group receiving mobile games in addition to the standard treatment will experience a better rehabilitation process in terms of thumb functionality, pain, and edema compared to the routine treatment group, and they will reach rehabilitation goals more quickly. Additionally, mobile games will increase motivation for home exercises and improve adherence. This study will be the first to examine the use of mobile games in thumb rehabilitation and their effect on adherence to home exercises. Researchers anticipate that the results of this study will inspire both clinicians and future research, reaching a wider audience through presentations and publications.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18-65
* With sufficient communication skills
* Experiencing pain and functional impairment in the thumb (e.g., thumb fractures, tendon injuries, nerve injuries, osteoarthritis, trigger thumb, carpal tunnel syndrome, ligament injuries, soft tissue damage, etc.),
* who are willing to volunteer.

Exclusion Criteria:

- Illiteracy, lack of a smartphone, or the presence of neurological, orthopedic, or rheumatological chronic diseases in the affected limb.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2024-05-15 (Actual); Primary Completion 2025-02-01 (Estimated); Study Completion 2025-02-01 (Estimated)

PRIMARY OUTCOMES:
The Quick Disabilities of the Arm, Shoulder, and Hand (Quick DASH) Questionnaire | 1st week and 4th week
  The Quick Disabilities of the Arm, Shoulder, and Hand (Quick DASH) is a valid and reliable scale consisting of 11 questions that assess the functional status and symptoms of the upper extremity in cases of disease and injury. It is a shorter version of the original DASH. Each question has five response options (1: no difficulty, 5: unable to do). To calculate the score, at least 10 questions must be answered. The total score is calculated out of 100 points, with higher scores indicating greater levels of disability.

SECONDARY OUTCOMES:
Duruöz Hand Index (DEİ) | 1st week and 4th week
  It is an 18-item scale that assesses hand function in activities such as cooking, dressing, personal hygiene, and other daily tasks, without inquiring about pain, numbness, social life, or psychological state. The assessment takes approximately three minutes to complete. The score is calculated out of 90 points, with higher scores indicating greater limitations and difficulty in daily living activities.
Assessment of Range of Motion (ROM) | 1st week and 4th week
  The most commonly used objective method for assessing joint motion in the literature is goniometric measurement, which is both valid and reliable. Although the universal goniometer is the most frequently used goniometric tool, the finger goniometer is also one of the types of goniometers. An appropriate, satisfactory, adaptable, and reliable goniometer tool should be selected based on the situation. Measuring joint motion is difficult due to the large number of joints, small area, and complex movements involved. Due to the inherent challenges of the hand, we will prefer the finger goniometer in our study and measure the active flexion and extension angles of the thumb's metacarpophalangeal and interphalangeal joints.
Pain Assessment | 1st week and 4th week
  Patients' pain during night, rest, and activity will be assessed using the Visual Analog Pain Scale (VAS). The VAS is a subjective evaluation method consisting of a horizontal or vertical 10 cm straight line. It corresponds to the expressions 0: no pain, 10: extreme/unbearable pain. The patient is asked to mark a point on the line according to the severity of their pain, considering these endpoints. The distance from the marked point to 0 is measured and recorded in centimeters.
Assessment of Adherence to Home Exercises | 1st, 2nd, 3rd and 4th week
  Patients will be provided with a home exercise tracking chart to monitor adherence to home exercises. In this chart, the relevant boxes will be marked each day the patient performs the home exercises over a period of 3 weeks.

OTHER OUTCOMES:
Case Follow-up Form | 1st week
  This form will collect information from patients, including age (year), height (cm), weight (kg), occupation, education level, dominant hand, injured hand, type of injury, smoking and alcohol use, comorbidities, details of any surgery performed on the hand, and medications used. Based on the randomization result, the patient's assigned group will be recorded in this form. The results of the range of motion measurements will also be entered into the table in this form. The Visual Analog Scale (VAS) (cm)will also be included in this form.

CONTACTS AND LOCATIONS:
Locations (1):
- Kırşehir Ahi Evran University, Kirşehi̇r, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No